CLINICAL TRIAL: NCT06190756
Title: Effect of Intra-cardiac Hydrostatic Pressure Gradient in Cardiac Filling and Ejection
Brief Title: Impact of Gravity on Cardiac Hemodynamics
Acronym: ACUITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: INSERM UMR-S 1075 COMETE, Caen, France (Unknown); CNRS UMR 5220 INSERM U1294 CREATIS ,Université Lyon 1, INSA Lyon, France (Unknown); Jozef Stefan Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-0077
Record Dates: First submitted 2023-11-23; First posted 2024-01-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Diabetes type1; Healthy
Keywords: Gravity; Intracardiac pressure gradients; Cardiac function; Echocardiography; Lower Body Negative Pressure; Tilt-test; Diabetes; Color Doppler M mode
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Circulation; Head-Down Tilt; Lower Body Negative Pressure

STUDY DESIGN:
Intervention Model Description: Comparison of two groups : Control vs. Diabetes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1 Diabetic group (Experimental): Group with diabetic patients
  Interventions: Other: Cardiovascular and Baroreflex stimulation by Tilting; Other: Cardiovascular and Baroreflex stimulation by Lower Body Negative Pressure
- Healthy Control Group (Other): Control group with healthy participants
  Interventions: Other: Cardiovascular and Baroreflex stimulation by Tilting; Other: Cardiovascular and Baroreflex stimulation by Lower Body Negative Pressure

INTERVENTIONS:
Other: Cardiovascular and Baroreflex stimulation by Tilting — Tilt of the patient at 4 angles (22°, 42°, 58° and 80°), the order is randomized for 3 angles (22°, 42°, 58°) while 80° will always be last.
  Other Names: Tilt
Other: Cardiovascular and Baroreflex stimulation by Lower Body Negative Pressure — The patient will undergo 4 level of LBNP (10Torr, 20Torr, 35Torr, 50Torr), the order is randomized for 3 intensities (10Torr, 20Torr, 35Torr) while 50Torr will always be last.
  Other Names: LBNP

SUMMARY:
The goal of this clinical trial is to define and compare pre-load dependance of the cardiac function according to the intracardiac hydrostatic gradient of pressure in healthy and diabetic populations.

Participants will undergo 4 tilt angle and 4 lower body negative pressure intensities during which cardiovascular data will be assessed and a transthoracic echography will be performed.

DETAILED DESCRIPTION:
Gravitational force affects both the cardiac mass and the thoracic compartment. However, few studies in humans have explored whether the relationship between cardiac function and load-dependence varies according to the orientation of the heart in space (e.g. between the upright and supine positions) and therefore according to gravitational stress.

Thirty-two volunteers (16 healthy subjects and 16 subjects with type I diabetes) will be included in the study. Each subject will be analysed over half a day in the Inserm COMETE laboratory. Measurements of the intra-cardiac hydrostatic pressure gradient (reflecting gravitational force) and indicators of cardiac function will be analysed by transthoracic echocardiography using dedicated post-processing software. These measurements will be compared at identical pre-load on the basis of the relationship between thoracic impedance and angle of vertical inclination using a Tilt Test on the one hand and between thoracic impedance and Lower Body Negative Pressure (LBNP) depression in the supine position on the other. In the supine position, the echocardiogram will be repeated for each subject with different levels of intensity of preload decrease by LBNP up to a maximum of -50 torr, and compared with different angles of vertical inclination head up up to +80° on the Tilt Test.

The study aims to compare the contribution of intra-cardiac hydrostatic force to cardiac filling and ejection mechanics in a population of healthy volunteers and subjects with diabetes.

The goal is to define and compare the pre-load dependence of the cardiac function indices studied according to the anatomical supine posture with zero intra-cardiac hydrostatic gradient with the standing posture during which the hydrostatic force is expressed between the cardiac base and apex. The hypothesis is that cardiac filling and ejection are improved when the longitudinal axis of the heart is anatomically oriented in the standing position compared with the supine position, by restoring the intraventricular hydrostatic pressure gradient. Comparing a group of healthy subjects with a group of subjects with diabetes will enable to assess whether the dependence of cardiac function on the orientation of the heart in space is more marked in the presence of subclinical impairment of myocardial function.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to the social security system
* Patient informed of the study and having signed an informed consent form
* Type 1 diabetes for at least 10 years followed at Caen University Hospital, equipped with a continous glucose monitoring system

Exclusion Criteria:

* Trained athletes (≥ 6 hours of sustained physical exercise >70% VO2max per week for > 6 months)
* Chronic cardiovascular disease or cardiovascular treatment
* Personal history of chemotherapy and/or thoracic radiotherapy
* Cerebral and/or spinal disease
* Inclusion of the subject in another biomedical research protocol of interventional type (during the study or in the 3 months prior to inclusion)
* Pregnant, breast-feeding or parturient women
* Adults under legal protection (guardianship, curators) or unable to express their consent or deprived of their freedom

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-06-22 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Heart rythme | baseline, during the intervention
  continuous electrocardiogram monitoring for assessing the variation of heart frequency
Arterial blood pressure | baseline, during the intervention
  continuous central arterial pressure monitoring using Finapress
thoracic Impedancemetry | baseline, during the intervention
  estimation of body fluid variation as a surrogate of prelaod
Echocardiography | baseline, during the intervention
  non invasive diastolic intraventricular pressure gradient

CONTACTS AND LOCATIONS:
Locations (1):
- Inserm 1075 Comete, Unicaen, Caen, France

IPD SHARING:
Plan to Share IPD: No